# Participant Name: Study Title: Randomized Trial of Titrated Disease Management for Patients With Hypertension Principal Investigator: Dr. George L. Jackson, PhD, MHA Research Informed Consent Form Version Date: 2014-08-25  VA Form 10-1086 Date: Study Title: Randomized Trial of Titrated Disease Management for Patients With Hypertension VAMC: Durham

Please read this form carefully. It tells you important information about a <u>voluntary</u> research study. As your study doctor or study staff discusses this consent form with you, please ask him/her to explain any words or information that you do not clearly understand. It is important that you understand the information on this form. If you would like to check that this study is approved by the Durham VAMC's Institutional Review Board, please call the research office at (919) 286-6926 or (888) 878-6890, extension 6926.

## WHY IS THIS RESEARCH BEING DONE?

The purpose of this research is to test ways to control blood pressure among veterans.

You are being asked to participate in this research study because you are a patient receiving primary care at the Durham Veterans Affairs Medical Center, including Veteran Affair Community Based Outpatient Clinics, are over the age of 18 and have or had uncontrolled high blood pressure. **We will enroll participants until we select up to 400 patients** for this study and will ask each enrolled participant to be in the study for **18 months**.

## What is the experimental part of this research study?

You will receive education about high blood pressure over the telephone from a Licensed Practical Nurse (LPN), Registered Nurse (RN), or a Pharmacist. Some patients will be asked to check their blood pressure at home and some patients will receive special review of any blood pressure medicines that they may be taking.

## WHAT PROCEDURES, DRUGS, OR TREATMENTS ARE INVOLVED IN THIS RESEARCH STUDY?

- This study involves four (4) in-person interviews (including today) and possibly one (1) audiorecorded phone interview for which we would call you towards the end of the study to see how you felt about your participation in this study.

## Baseline (first) Study Visit:

At the first visit, which is this visit today, I will take 3 blood pressure readings and measure your height and weight and pulse. If an error occurs we may retake your blood pressure up to a total of 6 readings. I will then ask you a set of questions about you and your health. The last step is that you will be assigned to one of two study groups using a procedure like drawing numbers from a hat. You will be told which group you have been assigned to. The investigator may end your participation in

| Subject Identification (last, first, middle) and Social Security Number: | Unstamped forms are invalid |
|---|---|
| | IRB Approved DVAMC Date 9/11/14 |



the study without regard to your consent for one or more of the following reasons: investigator decides that continuing you participation could be harmful to you, or failure to follow instructions of investigator and/or study staff.

For women who are pregnant or may become pregnant: If you are pregnant or plan to become pregnant in the next two years, you may not participate in this study because the drugs used to manage blood pressure may be different if you are pregnant. When you come in for your 6 and 12 month study visit, you will be asked if you are pregnant or plan to become pregnant. If you receive care from the study pharmacist, the pharmacist will ask if you are pregnant or plan to become pregnant before the end of the study. If the answer is yes, the investigator may end your participation in the study.

## STUDY GROUP 1: Adjusted Disease Management Group

If you are chosen for this group, we will use the blood pressure reading from today to assign you to receive either:

## 1. Monthly phone calls from a Registered Nurse (RN)

If you are in this group, you will get telephone calls approximately once a month about how to best manage your own blood pressure. You will also be asked to check your blood pressure at home and report the information to the RN. We will offer to get you a home blood pressure machine from the VA if you do not already have one. It is anticipated that these calls will last about 20 minutes. However, call length will depend on your individual needs. In order to allow us to see how well the RN is doing at providing you with the phone calls, we may record one or more calls so that senior study staff can listen to the quality of the phone calls. These recordings will only be accessed by authorized study staff.

## <u>OR</u>

## Monthly phone calls from a Pharmacist.

If you are in this group you will get telephone calls approximately once a month about how to best manage your own blood pressure. You will also be asked to check your blood pressure at home and report the information to the Pharmacist. We will get you a home blood pressure machine from the VA if you do not already have one. In addition, the pharmacist will review any blood pressure medicine you may be on. The pharmacist may make changes in these medicines. Your primary care doctor will be notified about any changes. It is anticipated that these calls will last about 30

Unstamped forms are invalid

IRB Approved

DVAMC
Date 9/11/19

# Participant Name: Study Title: Randomized Trial of Titrated Disease Management for Patients With Hypertension Principal Investigator: Dr. George L. Jackson, PhD, MHA Research Informed Consent Form Version Date: 2014-08-25  VA Form 10-1086 Date: Study Title: Randomized Trial of Titrated Disease Management for Patients With Hypertension VAMC: Durham

minutes. However, call length will depend on your individual needs. In order to allow us to see how well the pharmacist is doing at providing you with the phone calls, we may record one or more calls so that senior study staff can listen to the quality of the phone calls. These recordings will only be accessed by authorized study staff.

## 6 and 12 month readjustment of your disease management level:

After approximately 6 and 12 months at the study visits (described below) your blood pressure will be checked again. You might continue services from the same person (i.e. RN or Pharmacist). If you are getting phone calls from a nurse and your blood pressure control gets worse, you may then start getting calls from the pharmacist. If you are in the pharmacist group and your blood pressure improves, you may be switched to the registered nurse group.

If your blood pressure is in control during the time it is scheduled to be readjusted, you will be switched to a booster level group where you will get a call about how to manage your blood pressure approximately every two months from a licensed practical nurse (LPN) or similar member of the research team. It is anticipated that these calls will last about 10 minutes. However, call length will depend on your individual needs. In order to allow us to see how well the LPN is doing at providing you with the phone calls, we may record one or more calls so that senior study staff can listen to the quality of the phone calls. These recordings will only be accessed by authorized study staff.

## Automatically Receiving Disease Management Services From the Pharmacist:

You will be moved to the pharmacist group automatically in either of the following situations:

1. Your average home systolic blood pressure ("top number" of your blood pressure) is equal to or over 160 mmHg.

## <u>OR</u>

2. Your average systolic blood pressure ("top number" of your blood pressure) at a visit for this research study is equal to or over 160 mmHg.

## OR

3. You are hospitalized due to a heart attack (also called an MI or a myocardial infarction) and/or a stroke.

## STUDY GROUP 2 - Controlled Disease Management Group

Patients randomly assigned to this group will get a call about how to manage your blood pressure approximately every two months from a licensed practical nurse (LPN) or similar member of the

| Unstampe | ed forms are invalid |
|----------|----------------------|
| idB Ap | proved |
| DVAM | Ċ, F. |
| Date_ | 9/11/14 |

# Participant Name: Study Title: Randomized Trial of Titrated Disease Management for Patients With Hypertension Principal Investigator: Dr. George L. Jackson, PhD, MHA Research Informed Consent Form Version Date: 2014-08-25 IRB Template: 2014-06-12 VA Form 10-1086 VAMC: Durham

research team. It is anticipated that these calls will last about 10 minutes. However, call length will depend on your individual needs. In order to allow us to see how well the LPN is doing at providing you with the phone calls, we may record one or more calls so that senior study staff can listen to the quality of the phone calls. These recordings will only be accessed by authorized study staff.

## Study Visits for all participants:

## (6 month study visit, 12 month study visit, and 18 month study visit):

You will be asked to make 3 research visits after your baseline visit. These will be 6, 12, and 18 months after your baseline visit. At each of these visits, we will measure your blood pressure, height, weight and pulse. We will also ask you questions about your understanding of high blood pressure and changes in your weight, smoking status, regular use of medication and other lifestyle factors.

This visit should take no more than 60 minutes.

### Possible Audio Recorded Phone Interview:

It is possible that we may ask to speak with you towards the end of the study to find out how you felt about your participation in this study. This interview is optional. The questions we ask would focus on your opinion about different parts of the study. The conversation will be audio recorded on a VAowned computer. The conversation will be later written down using VA-owned computer software, and the recording will be destroyed.

This is an optional part of the study and you have the right to refuse to participate in it if asked. **This phone interview should take no more than 30 minutes.** Individuals participating in the telephone interview will not receive any payment for the telephone interview.

## WILL ANY OF MY DATA, BLOOD, TISSUE OR OTHER SAMPLES BE STORED AND USED FOR FUTURE RESEARCH?

## Use of Medical and Related Information:

To better understand the reason our study works (or doesn't work), or to understand other aspects of your health or healthcare that may lead to lower risk of heart disease, we will access medical information about you stored in VA medical or other records that provide information on your health, healthcare, or services received from the Department of Veterans Affairs. In addition, we may get similar information from Medicare or Medicaid records if you have either Medicare or Medicaid. Only authorized study staff members will be granted access to the data. Any data that could be used to identify you will be stored on secure computers managed by the Durham VA Medical Center.

| Unstamped forms are ir | valid |
|------------------------|-------|
| IRB Approved | |
| DVAMC<br>Date9// | |
| Date9/11/1 | 4 |

# Research Informed Consent Form Version Date: 2014-08-25  IRB Template: 2014-06-12 VA Form 10-1086 Participant Name: Date: Study Title: Randomized Trial of Titrated Disease Management for Patients With Hypertension Principal Investigator: Dr. George L. Jackson, PhD, MHA VAMC: Durham

## Future Use of Study Data:

We request to keep the data collected about you during this study on high blood pressure of veterans for use in future research. This includes, but is not necessarily limited to, seeing how your health and healthcare change after you have completed this study. There is the possibility that other researchers working on high blood pressure or other cardiovascular disease issues may request to use the information collected in this study to answer other research questions. We may also use information from your medical records described above to look at the long-term effect of our study procedures on your health and healthcare. Only authorized study staff members will be granted access to the data. Any data that could be used to identify you will continue to be stored on secure computers managed by the Durham VA Medical Center.

## CAN I REFUSE TO BE IN THIS RESEARCH STUDY OR WITHDRAW AT A LATER TIME?

Absolutely. You do not have to join this or any other research study. If you do join and later change your mind, you may quit at any time. If you withdraw from the study, no new data about you will be collected for study purposes. If you refuse to join or if you withdraw from the study, there will be no penalty or loss of any benefits to which you are otherwise entitled. This will not affect your relationship with or treatment by the Veterans Health Administration (VHA) or your rights as a VHA patient. You will still receive all the medical care and benefits for which you are otherwise eligible.

## WHAT OTHER OPTIONS DO I HAVE?

Taking part in this study is your choice. You have the option not to participate

## HOW LONG WILL I BE IN THIS RESEARCH STUDY?

Over the next 18 months this study will involve four (4) in-person interviews (including today) which may last approximately 45 – 90 minutes. Depending on which group you are assigned you will receive home telephone calls either every month or every other month and possibly which may last approximately 10 to 30 minutes each. We may ask you to participate in one (1) audio-recorded phone interview for which we would call you towards the end of the study to see how you felt about your participation in this study; time of this call will depend on your individual responses.

WHAT ARE THE RISKS AND DISCOMFORTS OF PARTICIPATING IN THIS RESEARCH STUDY?

| Unstamped forms are invalid |
|-----------------------------|
| IRB Approved |
| DVAMC<br>Date 9/11/14 |

# Participant Name: Research Informed Consent Form Version Date: 2014-08-25  IRB Template: 2014-06-12 VA Form 10-1086 Participant Name: Date: Study Title: Randomized Trial of Titrated Disease Management for Patients With Hypertension Principal Investigator: Dr. George L. Jackson, PhD, MHA VAMC: Durham

You may experience some pressure or feelings of discomfort during the blood pressure measurements. The study intervention is likely to encourage you to try new foods and increase exercise. This may lower blood sugar. You may have an allergy to a new food. Risks from increased physical activity will be minimized by encouraging moderate rather than vigorous activity. Most importantly, if the pharmacist changes your medications, you may experience side effects from those medications and from the lowering of your blood pressure and blood sugar.

Also, some of the questions we ask during the survey may be considered sensitive to some people; we will skip any question that you do not want to answer. All surveys are kept confidential. All efforts will be taken to ensure that your information will be kept confidential. No additional risks to you are anticipated. If you experience discomfort that you think may be related to the research, you can call the study team.

## WILL I BENEFIT FROM TAKING PART IN THIS RESEARCH STUDY?

You may not personally be helped by taking part in this study, but your participation may lead to knowledge that will help others. You may see possible improvements in your health and in your health education.

## DOES PARTICIPATION IN THIS RESEARCH STUDY COST ANYTHING?

There will be no costs to you for any of the research treatment or research testing done as part of this research study. Some Veterans are required to pay co-payments for medical care and services provided by VA. These co-payment requirements will continue to apply to medical care and services provided by VA that are not part of this study.

## WILL I RECEIVE ANY COMPENSATION (MONEY OR OTHER) FOR TAKING PART IN THIS RESEARCH STUDY?

You will be responsible travel costs to the visits; travel vouchers cannot be provided for research-only visits. You will be paid \$15 for completing each of the four in-person visits. Therefore, the maximum compensation for participating in this study is \$60. This payment will come by a method determined by VA policy and may be cash reimbursement, electronic fund transfer, a VA check, or another form of VA payment.

Unstamped forms are invalid

IRB Approved
DVAMC
Date 9/11/14



## ARE THERE REASONS THAT MY RESEARCH PARTICIPATION MAY END EARLY?

Dr. George L. Jackson may take you out of the study without your consent for one or more of the following reasons: ... investigator decides that continuing you participation could be harmful to you, or failure to follow instructions of investigator and/or study staff.

For women who are pregnant or may become pregnant: If you are pregnant or plan to become pregnant in the next two years, you may not participate in this study because the drugs used to manage blood pressure may be different if you are pregnant. When you come in for your 6 and 12 month study visit, you will be asked if you are pregnant or plan to become pregnant. If you receive care from the study pharmacist, the pharmacist will ask if you are pregnant or plan to become pregnant before the end of the study. If the answer is yes, the investigator may end your participation in the study.

## WHAT WILL HAPPEN IF I AM INJURED WHILE PARTICIPATING IN THE RESEARCH STUDY?

The VA will provide necessary medical treatment should you be injured by being in this study. You will be treated for the injury at no cost to you. This care may be provided by the Durham VAMC or arrangements may be made for contracted care at another facility. No promises have been given to you as the results and the risks of a research study are not always known in advance. Every reasonable safety measure will be taken to protect your well-being. You have not released this institution from liability for negligence. In case of research related injury resulting from this study, you should contact your study team. If you have questions about compensation and medical treatment for any study related injuries, you can call the medical administration service at this VA Medical Center at 919-286-6957.

## WILL MY CLINICAL OR OTHER RESEARCH TEST RESULTS BE SHARED WITH ME?

We will let you and your physician know of any important discoveries made during this study which may affect you, your condition, or your willingness to participate in this study.

## WILL THE RESULTS OF THIS RESEARCH STUDY BE SHARED WITH ME?

We do not plan to share research study results.

| unstamped to | orms are invalid |
|------------------------|------------------|
| IRB Approv | ved |
| DVAMC<br>Date <b>9</b> | 11/11 |



## DO ANY OF THE RESEARCHERS HAVE A FINANCIAL INTEREST RELATED TO THIS RESEARCH STUDY?

This study is sponsored by a grant from VA Health Services Research & Development. Portions of Dr. George Jackson's, the principal investigator of the study, and his research team's salaries are paid by this grant.

## HOW WILL MY RESEARCH DATA BE PROTECTED AND SECURED?

There are VA rules (called records control requirements) about how long your research records are kept. Right now the rules say your research records cannot be destroyed. This may change in the future; at that time we will follow the new VA rules. Your medical records will be maintained according to this medical center's requirements. All research records, including survey and audio files, will be in the care of Dr. Jackson. They will be safeguarded under lock and key at locations managed by the Durham VA Medical Center. Study data storage will involve computer files that will be password protected. Files containing names and addresses will have a separate password and will be accessible only to personnel who need to contact subjects. All survey data will be obtained using a VA owned computer that is connected to the Durham VAMC computer network. If the computer network is not available, survey data may be obtained using an encrypted VA owned computer or by paper surveys. To provide the greatest assurance possible that accidental disclosure will NOT take place, data files not directly needed to conduct the study are organized by study ID number and have no names or other identification attached. All databases are secured with password protection to prevent unauthorized access and paper copies of information are kept in locked file cabinets. The paper research records will be shredded and information in the electronic format will be deleted or purged from data files; both are in accordance with the VA record control requirements for destruction of sensitive information.

## WILL ANYONE ELSE HAVE ACCESS TO MY RESEARCH DATA?

If results of this study are reported to others, you will not be identified by name, by recognizable photograph, or by any other means without your specific consent.

Your research records may be reviewed by Durham VA staff who are responsible for the safe conduct of this research. We may also provide your research records to federal agencies such as the Office for Human Research Protections (OHRP), the VA Office of the Inspector General (OIG), and the Office of Research Oversight (ORO). We will not share any information with these groups outside the VHA

| Unstampe | ed forms are invalid |
|----------|----------------------|
| IRB Ap | proved |
| DVAM | |
| Date_ | 9/11/14 |

# Research Informed Consent Form Version Date: 2014-08-25  IRB Template: 2014-06-12 VA Form 10-1086 Participant Name: Study Title: Randomized Trial of Titrated Disease Management for Patients With Hypertension Principal Investigator: Dr. George L. Jackson, PhD, MHA VAMC: Durham

unless they agree to keep the information confidential and use it only for the purposes related to the study. Any information shared with these outside groups may no longer be protected under federal law. These groups may disclose your information to other groups. If the sponsor receives identified information, it is then the sponsor, and not the VA, who is responsible for the security of the information.

## WHO DO I CONTACT IF I HAVE QUESTIONS OR CONCERNS ABOUT THE RESEARCH STUDY?

If you have questions about the research or need to talk to the study team, you can contact the principal investigator at (919) 286-6936 during the day and at (919) 210-6468 after hours. If you have questions about the research or your rights as a research participant, would like to obtain information, offer input, or have other concerns or complaints, you may contact the administrative officer of the research service at (919) 286-0411, extension 7632.

## **AFFIRMATION FROM PARTICIPANT**

My rights as a research participant have been explained to me, and I voluntarily consent to participate in this study. I have received an explanation of what the study is about and how and why it is being done. I authorize the use and disclosure of my identifiable information as described in this form. I will receive a signed copy of this consent form. If I am a VA patient, a copy of this consent form will be placed in my medical record.

| Participant's Signature/Legally Authorized Representative* | Date |
|------------------------------------------------------------|------|
| Signature of Investigator or Person Obtaining Consent | Date |

Unstamped forms are invalid
IRB Approved
DVAMC
Date 9/11/14

| Department of Veterans Affairs | HIPAA Authorization for Release of Protected<br>Health Information for Research Purposes | |
|---|---|---|
| Title of Study: Randomized Trial of Titrated Disease Management for | | Version Date: 5/29//2012 |
| Patients with Hypertension | | |
| Principal Investigator: George L. Jackson, Ph.D. | . MHA | VAMC: Durham |

You have been asked to participate in a research study under the direction of George L. Jackson, Ph.D., MHA and *his* research team. The purpose of this study is to improve the health of veterans with high blood pressure.

By signing this document, you will authorize the Veterans Health Administration (VHA) to provide *George L. Jackson* and *his* research team the authority to use and disclose the following information about you:

**Prior or Future Demographic information:** name, race, gender, age, home address, phone numbers, information necessary to enable you to receive electronic fund transfers including possibly bank account information and other information that the Department of Veterans Affairs or the Veterans Health Administration maintains about your background or identity.

**Prior or Future Medical Information:** prior and future blood pressure readings (systolic and diastolic), prior and future healthcare visits, prior and future prescriptions, cardiovascular diagnosis/other diagnoses, pregnancy, height, weight, and other health or healthcare information maintained by the Department of Veterans Affairs or the Veterans Health Administration.

**Prior or Future Laboratory values**: glycosylated hemoglobin (A1C), cholesterol, low density lipoprotein (LDL), high density lipoprotein (HDL), thyroid panel, liver enzyme. potassium, creatinine, or other prior or current laboratory values maintained by the Department of Veterans Affairs or the Veterans Health Administration.

Survey information: surveys to include audio recordings.

Automated VA Form 10-0114

The information collected also may possibly include the following health conditions: substance abuse problems [ X ] HIV [ X ] AIDS [ X ] mental health conditions [ X ] sickle cell anemia [ X ]

**Medicare or Medicaid Record Information:** If you have health coverage through Medicare or Medicaid, prior or future information on health or healthcare services recorded by Medicare or Medicaid may be obtained.

You do not have to sign this Authorization. If you decide not to sign the Authorization:

- It will not affect your regular medical care and rights as a VHA patient.
- You will not be allowed to participate in this research study.

| IMPRINT PATIENT DATA CARD | APPROVED |
|---------------------------|----------|
| | 3/13/17 |

| Department of Veterans Affairs | HIPAA Authorization for Release of Protected Health Information for Research Purposes | |
|---|---|---|
| Title of Study: Randomized Trial of Titrated Disease Management for | | Version Date: 5/29//2012 |
| Patients with Hypertension | | |
| Principal Investigator: George L. Jackson, Ph.D. | , MHA | VAMC: Durham |

This authorization will expire when this research study is closed with the Durham VA Medical Center Institutional Review Board.

You can withdraw this authorization at any time. To withdraw your authorization, you can write to Dr. Jackson at Durham VAMC, HSRD (152), 508 Fulton St, Durham NC 27705 or you can ask a member of the research team to give you a form to withdraw the authorization. If you withdraw this authorization, you will not be able to continue to participate in the study. This will not affect your rights as a VHA patient.

If you withdraw this authorization, Dr. George L. Jackson and his research team can continue to use information about you that has been collected. No information will be collected after you withdraw the authorization.

As part of the study, we may disclose your information and medical and/or research records to the Office for Human Research Protections (OHRP), the VA Office of the Inspector General (OIG), other government agencies, the Office of Research Oversight (ORO), the Durham VAMC Institutional Review Board (IRB), and/or local Research Compliance Officers. We will not share any information with these groups outside the VHA unless they agree to keep the information confidential and use it only for the purposes related to the study. Any information shared with these outside groups may no longer be protected under federal law. If the sponsor receives identified information, it is then the sponsor, and not the VA, who is responsible for the security of the information.

While this study is being conducted, you will not be allowed to see research-related medical records about you that are created or obtained by the research team. You may request to see the research-related medical records when the study is completed. This will not affect your doctor's ability to see your records as part of your normal health care.

The VHA complies with the requirements of the Health Insurance Portability and Accountability Act of 1996 and its privacy regulations and all other applicable laws that protect your privacy. We will protect your information according to these laws. Despite these protections, there is a possibility that your information could be used or disclosed in a way that it will no longer be protected. Our Notice of Privacy Practices (a separate document) provides more information on how we protect your information. If you do not have a copy of the Notice, the research team will provide one to you.

I have read this authorization form and have been given the opportunity to ask questions. If I have questions later, I understand I can contact **Dr. Jackson at 919-286-6936**. I will be given a signed copy of this authorization form for my records. I authorize the use and disclosure of my identifiable information as described in this form.

| Department of Veterans Affairs | HIPAA Authorization for Release of Protected<br>Health Information for Research Purposes | |
|---|---|---|
| Title of Study: Randomized Trial of Titrated Disease Management for | | Version Date: 5/29//2012 |
| Patients with Hypertension | | |
| Principal Investigator: George L. Jackson, Ph.D. | , MHA | VAMC: Durham |

The Paperwork Reduction Act of 1995 requires us to notify you that this information collection is in accordance with the clearance requirements of section 3507 of the Act. We may not conduct or sponsor, and you are not required to respond to, a collection of information unless it displays a valid OMB number. We expect that the time expended by all individuals completing this form will average 2 minutes. This includes the time to read the instructions, gather the necessary facts and fill out the form. The purpose of this form is to specifically outline the circumstances under which we may disclose data.

The execution of this form does not authorize the release of information other than that specifically described. The information requested on this form is solicited under Title 38, U.S.C. The form authorizes release of information that you specify in accordance with the Health Insurance Portability and Accountability Act, 45 CFR Parts 160 and 164, 5 U.S.C. 552a, and 38 U.S.C. 5701 and 7332. Your disclosure of information requested on this form is voluntary. However if the information, including Social Security Number (SSN) (the SSN will be used to locate records for release) is not furnished completely and accurately, Department of Veterans Affairs will be unable to comply with the request.

| SIGNATURE OF PARTICIPANT | Full SSN | DATE |
|--------------------------|----------|------|